CLINICAL TRIAL: NCT04569877
Title: Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) Inhalation to Prevent ARDS in COVID-19 Pneumonia (GI-COVID)
Brief Title: GM-CSF Inhalation to Prevent ARDS in COVID-19 Pneumonia
Acronym: GI-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KKS-279; 2020-001654-21 (EudraCT Number)
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-06

CONDITIONS: Severe Acute Respiratory Syndrome (SARS) Pneumonia; COVID-19 Pneumonia
Keywords: GM-CSF; COVID-19; ARDS
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molgramostim nebuliser solution (Experimental): 300μg molgramostim nebuliser solution
  Interventions: Drug: Molgramostim nebuliser solution
- Placebo nebuliser solution (Placebo Comparator): Placebo nebuliser solution
  Interventions: Other: Placebo nebuliser solution

INTERVENTIONS:
Drug: Molgramostim nebuliser solution — 300μg molgramostim nebuliser solution nebulised seven times within 7 days via rapid nebuliser system
  Arms: Molgramostim nebuliser solution
Other: Placebo nebuliser solution — Placebo nebulised seven times within 7 days via rapid nebuliser system
  Arms: Placebo nebuliser solution

SUMMARY:
To assess the safety and tolerability of inhaled molgramostim nebuliser solution in patients with COVID-19 pneumonia.

DETAILED DESCRIPTION:
COVID-19 pneumonia is induced by the newly emerging pandemic Severe acute respiratory Syndrome (SARS) coronavirus 2 and results in progression to the acute respiratory distress syndrome (ARDS). Apart from protective ventilation, fluid restriction, prone positioning and extracorporeal membrane oxygenation (ECMO), no specific therapeutic options exist to treat this devastating disease with a mortality rate of up to 50%. The growth factor granulocyte-macrophage colony-stimulating factor (GM-CSF) is widely recognized to promote differentiation and mobilization of different myeloid leukocyte subsets including neutrophils, tissue macrophages/dendritic cells or their circulating precursors. GM-CSF was found to be crucial for alveolar epithelial repair following hyperoxic and inflammatory lung injury.The aim of the current trial is to prevent progression to ARDS in COVID-19 pneumonia patients by preemptive GM-CSF Inhalation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form by the patient according to local regulations
2. Man or non-pregnant woman
3. Age ≥18 years
4. Willingness of patients with reproductive potential to use highly effective contraceptive methods by practicing abstinence or by using at least two methods of birth control from the date of consent to the end of the study. If abstinence could not be practiced, a combination of hormonal contraceptive (oral, injectable, or implants) and a barrier method (condom, diaphragm with a vaginal spermicidal agent) has to be used *.
5. Lab-confirmed COVID-19 pneumonia where pneumonia is diagnosed by radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR clinical assessment (evidence of rales/crackles on exam) AND pulse oximeter oxygen saturation ≤ 94% at room air in patients that do not have chronic hypoxia; or less than their baseline oxygenation in patients that suffer from chronic hypoxia
6. Negative serum pregnancy test in women of childbearing potentia

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Autoimmune thrombocytopenia, myelodysplastic syndromes with > 20% marrow blast cells
3. History or presence of hypersensitivity or idiosyncratic reaction to molgramostim (e.g. Leucomax®) or to related compounds (e.g. Leukine®)
4. Patient not able to use nebulizer device as well as immediately foreseeable mechanical ventilation of the patient
5. Simultaneous participation in another clinical trial with an experimental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation | During 15 days
  Need for mechanical ventilation within 15 days after randomization

SECONDARY OUTCOMES:
Clinical status of subject at day 15 and day 29 (on a 7-point ordinal scale): | At day 15 and day 29
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | At day 0 (day before first dose), day 1-9, and day 15
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] will be measured at day 0 (day before first dose), day 1-9, and day 15
Oxygen supply | At day 0, day 1-7, day 8-9 (24 hours/48 hours post dose) and day 15
  Need for oxygen supply (l/min) to reach peripheral oxygen saturation of 98%
Clinical parameter: temperature | Max. 48 hours before day 0, at day 0, day 1-7, day 8-9 and day 15
  Clinical parameter (4 times daily): temperature (°C degree)
Clinical parameter: blood pressure | Max. 48 hours before day 0, at day 0, day 1-7, day 8-9 and day 15
  Clinical parameter (4 times daily): blood pressure (mmHg)
Clinical parameter: heart beat | Max. 48 hours before day 0, at day 0, day 1-7, day 8-9 and day 15
  Clinical parameter (4 times daily): hear beat (beats per minute)
Clinical parameter: respiratory rate | Max. 48 hours before day 0, at day 0, day 1-7, day 8-9 and day 15
  Clinical parameter (4 times daily): respiratory rate (breaths per minute)
Severe acute respiratory syndrome coronavirus 2 polymerase chain reaction (PCR) | Max. 48 hours before day 0 and at day 8-9
  Presence of Severe acute respiratory syndrome coronavirus 2 nucleic acid by PCR test in swabs or tracheal aspirates/bronchoalveolar lavage
Laboratory: C-reactive protein test | At day 0, day 1-7, day 8-9 and day 15
  C-reactive protein test measures the amount of C-reactive protein in blood (mg/L)
Laboratory: ferritin | At day 0, day 1-7, day 8-9 and day 15
  Ferritin test measures the amount of ferritin in the blood (ng/ml)
Laboratory: Interleukin-6 | At day 0, day 1-7, day 8-9 and day 15
  Interleukin-6 test (IL-6) measures the amount of IL-6 in the blood (pg/ml)
Laboratory: procalcitonin | At day 0, day 1-7, day 8-9 and day 15
  Procalcitonin (PCT) test measures the amount of PCT in the blood in (μg/l)
Bacterial pneumonia | At day 0, day 1-7, day 8-9 and day 15
  Occurrence of secondary bacterial pneumonia
Vaso-active drugs | At day 29
  Days on vaso-active drugs in a 29-day period
Mortality | At day 29
  All-cause mortality
GM-CSF | At day 0 and day 1-7
  GM-CSF levels in serum

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Herold, Prof. Dr., Principal Investigator — Universitätsklinikum Giessen und Marburg (UKGM)
Locations (9):
- Germany (9):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Giessen und Marburg GmbH, Standort Giessen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Sana Klinikum Offenbach, Offenbach

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be provided after publication
Supporting Information: Study Protocol
Time Frame: 3 Months after publication
Access Criteria: Central server

REFERENCES:
- [Background] Arndt CA, Koshkina NV, Inwards CY, Hawkins DS, Krailo MD, Villaluna D, Anderson PM, Goorin AM, Blakely ML, Bernstein M, Bell SA, Ray K, Grendahl DC, Marina N, Kleinerman ES. Inhaled granulocyte-macrophage colony stimulating factor for first pulmonary recurrence of osteosarcoma: effects on disease-free survival and immunomodulation. a report from the Children's Oncology Group. Clin Cancer Res. 2010 Aug 1;16(15):4024-30. doi: 10.1158/1078-0432.CCR-10-0662. Epub 2010 Jun 24. PMID 20576718
- [Background] Ballinger MN, Paine R 3rd, Serezani CH, Aronoff DM, Choi ES, Standiford TJ, Toews GB, Moore BB. Role of granulocyte macrophage colony-stimulating factor during gram-negative lung infection with Pseudomonas aeruginosa. Am J Respir Cell Mol Biol. 2006 Jun;34(6):766-74. doi: 10.1165/rcmb.2005-0246OC. Epub 2006 Feb 10. PMID 16474098
- [Background] Cakarova L, Marsh LM, Wilhelm J, Mayer K, Grimminger F, Seeger W, Lohmeyer J, Herold S. Macrophage tumor necrosis factor-alpha induces epithelial expression of granulocyte-macrophage colony-stimulating factor: impact on alveolar epithelial repair. Am J Respir Crit Care Med. 2009 Sep 15;180(6):521-32. doi: 10.1164/rccm.200812-1837OC. Epub 2009 Jul 9. PMID 19590023
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Hamilton JA. Colony-stimulating factors in inflammation and autoimmunity. Nat Rev Immunol. 2008 Jul;8(7):533-44. doi: 10.1038/nri2356. PMID 18551128
- [Background] Herold S, Hoegner K, Vadasz I, Gessler T, Wilhelm J, Mayer K, Morty RE, Walmrath HD, Seeger W, Lohmeyer J. Inhaled granulocyte/macrophage colony-stimulating factor as treatment of pneumonia-associated acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Mar 1;189(5):609-11. doi: 10.1164/rccm.201311-2041LE. No abstract available. PMID 24579839
- [Background] Huang FF, Barnes PF, Feng Y, Donis R, Chroneos ZC, Idell S, Allen T, Perez DR, Whitsett JA, Dunussi-Joannopoulos K, Shams H. GM-CSF in the lung protects against lethal influenza infection. Am J Respir Crit Care Med. 2011 Jul 15;184(2):259-68. doi: 10.1164/rccm.201012-2036OC. Epub 2011 Apr 7. PMID 21474645
- [Background] LeVine AM, Reed JA, Kurak KE, Cianciolo E, Whitsett JA. GM-CSF-deficient mice are susceptible to pulmonary group B streptococcal infection. J Clin Invest. 1999 Feb;103(4):563-9. doi: 10.1172/JCI5212. PMID 10021465
- [Background] Matute-Bello G, Liles WC, Radella F 2nd, Steinberg KP, Ruzinski JT, Hudson LD, Martin TR. Modulation of neutrophil apoptosis by granulocyte colony-stimulating factor and granulocyte/macrophage colony-stimulating factor during the course of acute respiratory distress syndrome. Crit Care Med. 2000 Jan;28(1):1-7. doi: 10.1097/00003246-200001000-00001. PMID 10667491
- [Background] Papiris SA, Tsirigotis P, Kolilekas L, Papadaki G, Papaioannou AI, Triantafillidou C, Papaporfyriou A, Karakatsani A, Kagouridis K, Griese M, Manali ED. Long-term inhaled granulocyte macrophage-colony-stimulating factor in autoimmune pulmonary alveolar proteinosis: effectiveness, safety, and lowest effective dose. Clin Drug Investig. 2014 Aug;34(8):553-64. doi: 10.1007/s40261-014-0208-z. PMID 24890235
- [Background] Presneill JJ, Harris T, Stewart AG, Cade JF, Wilson JW. A randomized phase II trial of granulocyte-macrophage colony-stimulating factor therapy in severe sepsis with respiratory dysfunction. Am J Respir Crit Care Med. 2002 Jul 15;166(2):138-43. doi: 10.1164/rccm.2009005. PMID 12119223